CLINICAL TRIAL: NCT06672718
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of SPY002-091 in Healthy Participants
Brief Title: A Study of SPY002-091 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Spyre Therapeutics, Inc. (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPY002-091-101
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAD Cohorts, Experimental Arm (Experimental): Participants will receive a single dose of SPY002-091 in a dose escalation format
  Interventions: Drug: SPY002-091
- SAD Cohorts, Placebo Arm (Placebo Comparator): Participants will receive a single dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SPY002-091 — Experimental
  Other Names: SPY002
  Arms: SAD Cohorts, Experimental Arm
Other: Placebo — Placebo
  Arms: SAD Cohorts, Placebo Arm

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single- dose, first in human safety, tolerability, and pharmacokinetic study of SPY002-091 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Willing and able to attend the necessary visits to the CRU, comply with all testing requirements, remain at the study site unit for the duration of the confinement period and return for the outpatient visits

Exclusion Criteria:

* Participation in more than one cohort
* Evidence of clinically significant abnormality or disease
* Known history of illicit drug use or drug abuse, harmful alcohol use or alcoholism, and/or smoking or nicotine-containing product use within 3 months prior to the first dose of study drug
* History of severe allergic reactions or hypersensitivity
* Donation or loss of >1 unit of whole blood within 1 month prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | Up to 40 weeks
  Incidence, severity, and causal relationship of TEAEs

SECONDARY OUTCOMES:
Cmax | Up to 40 weeks
  Maximum concentration after single ascending doses
Tmax | Up to 40 weeks
  Time to reach maximum concentration after single ascending doses
AUC | Up to 40 weeks
  Area under the curve after single ascending doses
t1/2 | Up to 40 weeks
  Half life after single ascending doses
ADA | Up to 40 weeks
  Incidence of anti-drug antibody after single ascending doses

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Friedman, MD, Study Chair — Spyre Therapeutics
Locations (1):
- Spyre Site 1, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No